CLINICAL TRIAL: NCT03334994
Title: Facial Gingival Level Evaluation Following Soft Tissue Augmentation Using Connective Tissue Graft Around Immediate Dental Implants Versus Immediate Dental Implants Alone in the Esthetic Zone. Randomized Controlled Trial.
Brief Title: Facial Gingival Level Evaluation Following Soft Tissue Augmentation Using CTG Around Immediate Dental Implants vs Immediate Dental Implants Alone in the Esthetic Zone.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Parryhan Mohamed Abdelsamie, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 302017
Record Dates: First submitted 2017-11-02; First posted 2017-11-07 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Immediate Dental Implants Connective Tissue Graft Esthetic Zone
Keywords: Immediate dental implant, Connective tissue graft, Esthetic zone.

STUDY DESIGN:
Intervention Model Description: The patients was randomly classified into two groups:
  Group A: Patient will be treated with immediate implant alone. Group B: Patients will be treated with connective tissue graft combined with immediate implant.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinded participants: patient will be ensured by masking the instruments during the surgery. The patient will be informed of the steps of the surgery (as mentioned in the consent form) without getting into details. Blinding to the clinical, radiographic assessors is done by not involving them in sequence generation or allocation concealment or surgery performing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: immediate implant alone (Active Comparator): Patient will be treated with immediate implant alone.
  Interventions: Procedure: Intervention group:(Group B) connective tissue graft combined with immediate implant.
- (Group A) immediate implant alone (Active Comparator): Patient will be treated with immediate implant alone.
  Interventions: Procedure: Intervention group:(Group B) connective tissue graft combined with immediate implant.

INTERVENTIONS:
Procedure: Intervention group:(Group B) connective tissue graft combined with immediate implant. — Patients will be treated with connective tissue graft combined with immediate implant.

SUMMARY:
Aim of current study to evaluate connective tissue graft combined with immediate implant placement as an innovative option for less facial gingival tissue recession, less pocket depth and less clinical attachment loss versus immediate implant alone.

DETAILED DESCRIPTION:
P: Adult patients with single or multiple non-restorable teeth in esthetic zone I: Immediate implant + Connective tissue graft. C: Immediate implant alone. O: Primary Outcome: Facial gingival level Secondary Outcome: Patient satisfaction, probing depth, probing attachment loss, tissue biotype, keratinized mucosal width and bleeding on probing.

P.M will select patients from the outpatient clinic of the Oral Medicine and Periodontology Department - Cairo University. Screening of patients will continue until the target population is achieved. Identifying and recruiting potential subjects is achieved through patient database.

ELIGIBILITY:
Inclusion Criteria:

1. 18-55
2. Patients with single or multiple non-restorable teeth in maxillary anterior or premolar area.
3. Patients with adequate bone volume for the dental implant procedure.
4. Patients who are compliant to oral hygiene measures.
5. Patient consent approval and signing.

Exclusion Criteria:

1. Heavy smokers.
2. Systemic disease that contraindicates implant placement or surgical procedures.
3. No or poor patient's compliance.
4. Psychological problems.
5. Pathology at the site of intervention.
6. Pregnancy females.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Facial gingival level | Up to 6 months
  FGL was evaluated by measuring the distance between the level of soft tissues and the lower border of the customized template that was used as a reference line at three readings mesially, mid-facially and distally.

SECONDARY OUTCOMES:
Pain score | Up to 12 days
  Visual analog scale was recorded every day for 12 days follow-up and the patient marks on the line the point they feel that it represents their response
Patient satisfaction | Up to 6 month
  Post-Surgical Patient Satisfaction Questionnaire (PSPSQ). The patient questionnaire evaluates patients' perception and subjective admiration of the final result of the treatment
Tissue biotype | Up to 6 months
  Thickness of the peri-implant mucosa around the implant
Pink esthetic score | Up to 6 months
  seven different variables: mesial papilla, distal papilla, facial soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture at the facial aspect of the implant site
Width of keratinized mucosa | Up to 6 months
  distance from the mucogingival junction (MGJ) to the gingival margin
Bleeding on probing | Up to 6 months
  Bleeding was provoked by sweeping the peri-implant mucosal sulcus using a periodontal probe.
Probing depth | Up to 6 months
  distance from the peri- implant mucosal margin to the bottom of the peri-implant sulcus
Probing attachment level | Up to 6 months
  distance from the base of the peri-implant sulcus to the implant shoulder using periodontal probe at four sites

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Faculty of Dentistry., Giza, Egypt

IPD SHARING:
Plan to Share IPD: No